CLINICAL TRIAL: NCT01708395
Title: IBD-OPERA Database: Inflammatory Bowel Disease - Outcomes, Preferences, Education, Resource Utilization, Assessment Database
Brief Title: IBD-OPERA Database, UC Protocol
Acronym: OPERA
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Janssen Services, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: REMICADEIBD4007
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Inflammatory Bowel Disease
Keywords: Ulcerative colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1: First 50 patients
- Cohort 2: 2nd group of 50 patients

SUMMARY:
The investigators believe that patients with ulcerative colitis are able to report details of their own medical history accurately and record changes in clinical status effectively over time. Using an internet-based database the investigators will ask patients to report their own disease history, and the investigators will compare their reports to the medical record.

ELIGIBILITY:
Inclusion Criteria:

* MD documented diagnosis of ulcerative colitis
* current of past prescription for anti-TNF medication
* at least 18 years of age
* access to medical records to verify information
* 20% of participants will be patients diagnosed within 1 year of inclusion

Exclusion Criteria:

* unwilling or unable to provide informed consent for study participation
* unable to access or use internet
* less than 18 years of age
* diagnosis of crohn's disease or IBD-U
* illiterate or does not possess minimum level of literacy required to complete questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults over 18 years of age
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-10; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Validity of patient self reporting | 12 months
  The validity of patient self report on details of their ulcerative colitis compared to chart review. Validity is defined as a match between patient self report and medical records.

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States